CLINICAL TRIAL: NCT01813266
Title: Prospective Cohort Study: To Provide Evidence & Guidance in Hepatitis C Virus Screening, Comparing the New Birth Cohort Recommendations From the CDC, Versus Classical Traditional Strategies With Established Risk Factors.
Acronym: TPEGHCVS
Status: Withdrawn | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: hepcvirusscreeningtrial
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis C Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Hepatitis C virues enzyme immunosorbent assay screening; if positivie follow up testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Usual practice in screening for Hepatitis C virus.: Three clinics in this group will use this approach.
- USPTF risk factors to screen for chronic HCV infection.: 3 internal medicine clinics will use this screening strategy.
- USPTF/CDC recommendations to screen for chronic HCV infection.: 3 internal medicine clinics.

SUMMARY:
Although infection with the hepatitis C virus (HCV) can result in acute hepatitis; it more commonly progresses to chronic hepatitis. The acute process is most often asymptomatic. Acute HCV typically leads to chronic infection. Chronic HCV infection is usually slowly progressive. Approximately 5 to 20 percent of chronically infected individuals develop cirrhosis over a 20-30 year period of time. Chronic HCV is the most common cause of chronic liver disease, cirrhosis, hepatocellular carcinoma, and the most frequent indication for liver transplantation in the United States.

Screening for chronic HCV infection is crucial because chronic HCV infection is often asymptomatic, effective treatment is available, and untreated disease carries a high risk of morbidity and mortality. Expert opinion, recommendations, and guidelines for HCV screening do not all agree. All guidelines recommend screening patients at increased risk for HCV (ie: typical risk factors). In 2012, the Centers for Disease Control and Prevention (CDC) recommended screening all persons born between 1945 and 1965. At least two studies suggest that screening persons born between 1945 and 1964 or 1946 to 1970, respectively, is cost-effective. The studies estimated that if patients found to be HCV positive were treated with pegylated interferon, ribavirin, and direct acting antiviral therapy (for patients with HCV genotype 1), it would cost $35,700 to 37,700 per quality adjusted life-year. Screening based upon a birth cohort in patients without risk factors may lead to more false positive results.

Currently only 1 % of patients in the birth cohort of 1945-1965 who cared for by Intermountain Healthcare providers have been screened. Ambulatory care physicians are not effectively screening patients. It is unclear whether screening based on risk factors alone versus screening based upon risk factors and birth cohort most effectively manages the burden of chronic HCV infection for patients managed by Intermountain Healthcare providers. It is possible that the Intermountain Healthcare population differs in risk from the U.S. population,making guideline application less certain.

A well-designed prospective cohort study is needed to understand the risks and benefits of different HCV screening strategies on diagnostic yield and clinical outcomes.

The investigators hypothesize that screening based on a person's history of risk factors will detect chronic HCV infection in 2.7 % of the population tested; this would be according to national average. The investigators further hypothesize that screening based on birth cohort and risk factors will identify roughly the same percentage in the tested population. The investigators anticipate usable data within three months which should give us data to describe and publish the effectiveness of different screening strategies.

The investigators will identify patients with chronic HCV infection through this initial study who now require treatment and management. The investigators believe this group could be followed inexpensively for clinical endpoints for many years. This would then definitively define the effectiveness of screening strategies based on good evidence. No study has evaluated clinical outcomes associated with the different screening strategies for chronic hepatitis c virus infection.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS (limit one page)

1. Compare yield of risk based versus risk based and birth cohort screening for hepatitis C virus as a function of number invited to screen. The control group will receive the routine care as delivered normally by local medical practice. This will be conducted in the Salt Lake Area.
2. Determine cost in each arm of hepatitis C virus screening strategy.
3. Assess patient history for unknown risk factors for infection with HCV.
4. Create a registry of HCV positive and HCV negative patients to follow in future studies to determine long term outcomes.

Outcome Measures:

1. Rate of positive screening for HCV in each group as a function of number invited to screen.
2. Rate of persistent HCV infection in screen-positive patients based on confirmatory testing.
3. Determine percentage Utah population that test positive for HCV as compared to national average.
4. Listing of risk factors for each patient and analysis of risk factor tools to discover new risk factors and causes.

B. BACKGROUND AND SIGNIFICANCE (Limit two pages)

There has been much published in regards to recommendations to screen patients for HCV. Much of the attention is due to new treatments. Specific antiviral treatments to genotype 1 of HCV have received much attention. The reported sustained viral response in HCV genotype 1 with these new agents have been impressive but currently at great expense(12). With these new advances it has become paramount to identify patients early to avoid great morbidity and early mortality.

There are also disparate recommendations on screening for HCV between the Centers for Disease Control and Prevention and the United States Preventive Task Force. The American Association for the Study of Liver Diseases has sided with the CDC. The CDC has a new birth cohort recommendation in addition to risk factor screening versus the USPTF recommendation to do screening based upon risk factors only.

Given conflicting guidelines, tailored evidence to provide guidance to Intermountain clinicians would be useful; especially as the Intermountain population may differ from the U.S. population in risk making application of national guidelines more uncertain. This study will delineate the most effective screening approach for the population served, identify the rates of false positive tests, and delineate the costs of the screening strategies as recommended.

Currently only one percent of patients in the birth cohort of 1945-1965 and cared for by Intermountain Healthcare providers have been screened. Ambulatory practitioners are not effectively screening patients or may not believe these patients to be at sufficient risk to merit screening. It is unclear whether screening based on risk factors alone, or screening based upon risk factors and birth cohort recommendations most effectively manages the burden of chronic HCV infection for patients managed by Intermountain Healthcare providers.

A well-designed prospective cohort study is needed to understand the risks and benefits of different HCV screening strategies on diagnostic yield and clinical outcomes (9).

We hypothesize that screening based on established risk factors will detect HCV 2.7 % of the population tested. We believe that adding the proposed birth cohort in addition to risk factors for screening will not increase the number of those we identify with chronic HCV.

Once we have generated a registry of patients through this Initial study we believe this group could be followed inexpensively for clinical endpoints for many years to come. We would have a group of newly diagnosed chronically infected patients with HCV, identified by the CDC and USPTF guidelines. We then could ensure evidence base HCV treatment and follow endpoints of chronic liver disease and its complications. We would then be able to know if screening for hepatitis C virus is beneficial to the patient we care for and cost effective.

We have 885,000 patients of intermountain healthcare born between 1945 and 1965. Only one percent of them have been screened for HCV. In those screened 11% had positive HCV tests. The national average is 2.7 percent. This is not based upon any clear screening program. We appear to be screening for hepatitis C well below the national average. The state of Utah Epidemilogist's data indicate that 1% of Utahns have hepatitis C.

If we tested per CDC recommendation we would expect to diagnose 20,000 additional patients with HCV. If each individual were screened and those who tested positively received liver biopsy and treatment we could expect this to cost the system close to 3 billion dollars.

In summary, it is likely that many people with chronic HCV have not been identified and treated. In this study, we will determine the effectiveness of each screening strategies. This will inform clinicians about how to screen know how to screen for chronic HCV based on evidence and not recommendations. Further as we follow the newly diagnosed patients we will determine if our screening was effective following our evidence based management. We will also be able to measure costs as opposed to just calculations based on quality of life year.

C. EXPERIMENTAL DESIGN AND METHODS (Limit five pages)

We have identified 9 internal medicine offices in the Salt Lake area. We will divide the clinics into three groups (three clinics per each group). We are currently performing a prestratification of the groups to make sure there isn't an age, sex, or racial divergency. Group 1 would be our control group. The providers at these facilities will perform any hepatitis C virus screening as they would normally. Group 2 would provide risk factor screening per USPTF guide lines. Group 3 would use the CDC's recent birth cohort recommendations in addition to risk factor screening. The only exclusion criteria is if the patient has a test positive for hepatitis C virus or they give a positive history regarding infection.

We would like to identify 2000 patients for each strategy in 3 months. We would do this by asking office manager and physicians of clinics to let their office staff give a screening strategy form to each patient and ask them to be a part of this study. We will create sheets the patients can complete while they are waiting for their appointment. The clinical staff would then be asked to interpret and order the appropriate testing.

We will place the strategy on a one sided sheet of paper that can be given to all internal medicine patients between the age of 18 and 75.

I have enlisted the help of Dr. Greg Elliott, Scott Stevens, and Scott Woller and others in an steering committee to offer expert advice and guidance.

Strategies:

1. Screen for hepatitis C as per regular practice as is occurring in their clinics currently.

   1. Form would ask them if they ever had been tested for Hepatitis C.
   2. The rest of screening would be left to the provider's discretion.
2. Screen for hepatitis C as per conventional risk factors:

   a. A sheet with these risk factors will be provided i. Those with a history of illicit injection drug use or intranasal cocaine use, even if only used once ii. Those who received clotting factors made before 1987 iii. Those who received blood/organs before July 1992 iv. Those who have been informed that they received blood from a donor who later tested positive for HCV v. Those who were ever on chronic hemodialysis vi. Those with evidence of liver disease (persistently elevated alanine aminotransferase [ALT] level) vii. Those infected with HIV viii. Children born to HCV-infected mothers. ix. Those with a needle stick injury or mucosal exposure to HCV-positive blood x. Those who are a current sexual partner of an HCV-infected person xi. Incarcerated individuals xii. Healthcare, emergency, and public safety workers after needle stick/mucosal exposure to HCV-positive blood xiii. Children born to HCV-positive women xiv. Are spouses or household contacts of HCV-infected patients

   Those with these risk factors will be tested for HCV, HBV, and HIV

   Investigative factors:
   * Recipients of transplanted tissue after 1992
   * Those with a history of tattooing, body piercing
   * Those with a history of sexually transmitted diseases or multiple sex partners
   * Long-term steady sexual partners of HCV-positive persons

   Any exposure you are concerned about:______________________________.
3. Screen for hepatitis C by conventional risk factors and new CDC birth cohort recommendations.

   1. Anyone born in the United States between 1945 and 1965
   2. Those with a history of illicit injection drug use or intranasal cocaine use, even if only used once
   3. Those who received clotting factors made before 1987
   4. Those who received blood/organs before July 1992
   5. Those who have been informed that they received blood from a donor who later tested positive for HCV
   6. Those who were ever on chronic hemodialysis
   7. Those with evidence of liver disease (persistently elevated alanine aminotransferase [ALT] level)
   8. Those infected with HIV
   9. Children born to HCV-infected mothers.
   10. Those with a needle stick injury or mucosal exposure to HCV-positive blood
   11. Those who are a current sexual partner of an HCV-infected person
   12. Incarcerated individuals
   13. Healthcare, emergency, and public safety workers after needle stick/mucosal exposure to HCV-positive blood
   14. Children born to HCV-positive women
   15. Are spouses or household contacts of HCV-infected patients

Investigative risk factors:

* Recipients of transplanted tissue after 1992
* Those with a history of tattooing, body piercing
* Those with a history of sexually transmitted diseases or multiple sex partners
* Long-term steady sexual partners of HCV-positive persons

Any exposure you are concerned about:______________________________.

Guidance for initial positive HCV screen:

All patients will be tested for HCV, HBV, and HIV if they have the above risk factors.

If patients are found to be Hepatitis C positive by EIA, a HCV RNA quantity (viral load) would be performed. If the HCV RNA is negative and EIA is +, will order a HCV RIBA. (not PCR); if RIBA is negative this indicates a false positive EIA test.

Those patients with positive results would be notified by their primary physicians. We would provide a decision tree for work up and treatment of a newly found infection. Patients can be referred to gastroenterologists, hepatologists, and primary care providers who treat chronic hepatitis C virus infection.

F. IMPACT (Limit one page)

Hepatitis C virus is the leading cause of chronic liver disease in the United States, and is the leading reason for liver transplantation. Recent advances, in treatment , have made Hepatitis C virus chronic infection curable for many patients. It is important to identify, treat, and attempt to cure these patients, many of whom don't know they are affected.

Recommendations have been made to try and accomplish this. There needs to be evidence to guide our screening and therapy. With this study we could provide evidence to Intermountain, Utah, and I believe the greater medical community. In a few months we could have data that is publishable having compared the screening recommendations for HCV. We would know which if any of the screening strategies are superior in identifying chronic HCV.

We would do a follow up study, hopefully with additional funding from an outside group, having identified new carriers of chronic Hepatitis C. We would provide current evidence based antiviral treatments that are available based on genotype. This would allow us to see the comparative progression of liver disease with its subsequent complications in the three screened groups. We could follow these groups for up to 20 years and have evidence that would guide screening and treatment for HCV.

ELIGIBILITY:
Inclusion Criteria:

* anyone between the ages of 18 and 75 years old.

Exclusion Criteria:

* anyone who gives a history of chronic Hepatitis C virus infection or who has had a positive lab result in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: residents of Salt Lake County, Utah with pre-stratification to equalized sex, age, and ethnic similarity.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
superiority of Hepatitis C virus screening between three different strategies as far as identifying those with chronic hepatitis C virus infection. | 3-4 months
  Compare yield of risk based versus risk based and birth cohort screening for hepatitis C virus as a function of number invited to screen. The control group will receive the routine care as delivered normally by local medical practice. This will be conducted in the Salt Lake Area.
Cost of testing of screening for HCV. | 3-4 months
  Measure the cost of screening testing for HCV and follow up testing.
Develop a registry of patients with chronic HCV infection to follow through treatment. | 3-4 months
  Have a registry of patients we can follow for long term outcome.

SECONDARY OUTCOMES:
Identify new risk factors for Chronic Hepatitis C virus infection. | 3-4 months
  In Screening for Hepatitis C virus infection we are going to ask some novel risk factors to see if we identify any new risk factors for those who test positive.

CONTACTS AND LOCATIONS:
Overall Officials: brian a clements, d.o., Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Southern WN, Drainoni ML, Smith BD, Christiansen CL, McKee D, Gifford AL, Weinbaum CM, Thompson D, Koppelman E, Maher S, Litwin AH. Hepatitis C testing practices and prevalence in a high-risk urban ambulatory care setting. J Viral Hepat. 2011 Jul;18(7):474-81. doi: 10.1111/j.1365-2893.2010.01327.x. Epub 2010 May 20. PMID 20497311
- [Result] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Result] Velazquez RF, Rodriguez M, Navascues CA, Linares A, Perez R, Sotorrios NG, Martinez I, Rodrigo L. Prospective analysis of risk factors for hepatocellular carcinoma in patients with liver cirrhosis. Hepatology. 2003 Mar;37(3):520-7. doi: 10.1053/jhep.2003.50093. PMID 12601348
- [Result] Roblin DW, Smith BD, Weinbaum CM, Sabin ME. HCV screening practices and prevalence in an MCO, 2000-2007. Am J Manag Care. 2011;17(8):548-55. PMID 21851142
- [Result] Sanyal AJ; Governing Board the Public Policy, Clinical Practice, Manpower committees of the AASLD. The Institute of Medicine report on viral hepatitis: a call to action. Hepatology. 2010 Mar;51(3):727-8. doi: 10.1002/hep.23583. No abstract available. PMID 20198626
- [Result] Smith BD, Morgan RL, Beckett GA, Falck-Ytter Y, Holtzman D, Teo CG, Jewett A, Baack B, Rein DB, Patel N, Alter M, Yartel A, Ward JW; Centers for Disease Control and Prevention. Recommendations for the identification of chronic hepatitis C virus infection among persons born during 1945-1965. MMWR Recomm Rep. 2012 Aug 17;61(RR-4):1-32. PMID 22895429
- [Result] Duncan CJ, Stewart E, Fox R. Improving targeted screening for hepatitis C in the UK. BMJ. 2012 Oct 3;345:e6525. doi: 10.1136/bmj.e6525. No abstract available. PMID 23034845
- [Result] Sroczynski G, Esteban E, Conrads-Frank A, Schwarzer R, Muhlberger N, Wright D, Zeuzem S, Siebert U. Long-term effectiveness and cost-effectiveness of screening for hepatitis C virus infection. Eur J Public Health. 2009 Jun;19(3):245-53. doi: 10.1093/eurpub/ckp001. Epub 2009 Feb 5. PMID 19196737
- [Result] Chou R, Cottrell EB, Wasson N, Rahman B, Guise JM. Screening for hepatitis C virus infection in adults: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 Jan 15;158(2):101-8. doi: 10.7326/0003-4819-158-2-201301150-00574. PMID 23183613
- [Result] Chou R, Hartung D, Rahman B, Wasson N, Cottrell EB, Fu R. Comparative effectiveness of antiviral treatment for hepatitis C virus infection in adults: a systematic review. Ann Intern Med. 2013 Jan 15;158(2):114-23. doi: 10.7326/0003-4819-158-2-201301150-00576. PMID 23437439